CLINICAL TRIAL: NCT05224635
Title: The PROspective Observational Vascular Injury Trial (PROOVIT)
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 062.TRA.2021.D
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Vascular Injury
MeSH Terms: conditions — Vascular System Injuries | interventions — SPEG protein, human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects presenting to the emergency room: Chart review will include subjects presenting to the emergency room from the 1st of November 2021 through 1st of July 2024.
  Interventions: Procedure: Vascular Injury

INTERVENTIONS:
Procedure: Vascular Injury — The Society of Vascular Surgery has established a robust vascular disease registry but this organization's focus is on vascular disease and lacks capture of the data points necessary to discern trauma-specific outcomes. Recent military experience from the United States and United Kingdom, including the Balad Vascular Registry and the Global War on Terror (GWOT) Vascular Registry have provided a contemporary assessment of wartime vascular injury, but again these studies have been retrospective case series and registry reviews. Furthermore, applications of lessons learned in wartime vascular injury do not completely translate to management in trauma centers in the United States.

SUMMARY:
Evidence suggests that the rate of treatable vascular injury is increasing due to improved pre-hospital strategies. The increased rate of vascular trauma occurs in an era of increased sub-specialization, shifting training paradigms and the emergence of endovascular therapies. These factors, in combination with the baseline complexity of vascular trauma, make it particularly important that the management of this injury pattern be evidence-based. However, because all forms and distributions of vascular injury represent only 4% to 9% of trauma admissions, meaningful study of one injury pattern, patient population, therapeutic or surveillance strategy is difficult at a single institution. Further complicating such efforts is the fact that vascular trauma is managed by a wide range of surgical and now endovascular specialists, further fragmenting even a busy trauma institution's experience with vascular injury.

DETAILED DESCRIPTION:
Several institutions and groups have contributed important insight into the understanding of vascular injury management. However, many of the studies have been single-institution, poorly powered and retrospective. The lack of evidence-based practice is even more concerning given the devastating consequences associated with mismanaged vascular trauma. In light of the stated challenges associated with single-institution study of this injury pattern, the logical method with which to proceed is a prospective, multicenter, observational trail. To date no such registries exists which would allow the prospective aggregation of larger amounts of data pertaining to all phases of vascular trauma management.

Contemporary experience confirms that the management of vascular injury is more complicated than in the past. A multitude of new or updated diagnostic technologies including computed tomography angiography (CTA), magnetic resonance angiography (MRA), duplex and arteriography now exist and are in various degrees of vogue. A damage control approach to vascular trauma is widely championed and includes options for the use of tourniquets, temporary vascular shunts and fasciotomies. Controversies regarding the definitive management of vascular trauma abound and include the advisability of open versus endovascular treatment, decisions about the type of vascular conduit and the utility of venous injury repair lo list a few. Recommendations for surveillance after vascular trauma may include the use of duplex ultrasound or CTA to confirm long-term patency as well as choices related to the use of long-term anti-thrombotic therapy. Finally, it is not uncommon for an institution to find itself facing many of these decision points in the most challenging of all scenarios, the extremes of age including pediatric vascular injury.

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients; defined by the American College of Surgeons as individuals age: ≥16 years

  * CT/CTA, duplex, angiographic or clinical/ operative diagnosis of vascular injury following trauma
  * Initial management at Methodist Dallas Medical Center

Exclusion Criteria:

* Age: < 16 years
* No diagnosis of vascular injury
* Prisoner
* Subject transferred from another medical facility

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: • Adult trauma patients; defined by the American College of Surgeons as individuals age: ≥16 years
Sampling Method: Non-Probability Sample
Enrollment: 5718 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
establish an aggregate database | the 1st of November 2021 through 1st of July 2024
  establish an aggregate database of information of vascular trauma measured by Injury Severity Score (ISS): (range 0-75)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Burris, M.D., Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No